CLINICAL TRIAL: NCT03355599
Title: Investigating the Benefits of a 3D Camera for Recording Healing Wound Dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH19655
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Chronic and Non-healing Wounds
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3d camera (Other): 3d camera
  Interventions: Other: 3d camera

INTERVENTIONS:
Other: 3d camera — 3 D camera and associated software that introduces measurement and monitoring of wounds as a specific intervention

SUMMARY:
The study will explore whether a 3D camera data can provide a more accurate baseline measurement (compared to 2D images with manual measurement) to support better clinical decision making in referrals to tissue viability.

DETAILED DESCRIPTION:
Chronic and non-healing wounds are a significant problem to manage in community and represent a significant workload in community nursing. The current management for non-healing wounds includes referral to the tissue viability service, using a 2 D photographic image with assessment information. This study will pilot the use of a 3 D camera and associated software that introduces measurement and monitoring of wounds as a specific intervention. The introduction of 3 D measurement and monitoring of wounds will be compared with usual care. With a target recruitment of 30 patients via tissue viability, the pilot will report on the feasibility of using this outcome measure and the effectiveness of monitoring on wound closure or improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a non-healing wound and be over 18 years of age the criteria for non-healing wounds is as per 5.1 on the community nursing referral criteria when considering referral of patients to tissue viability:

'would expect that the wounds are deteriorating, chronic, non-healing or static or there are problems with the dressing regime'

Patients must be willing to provide written informed consent

Patients must have a registered Sheffield General Practitioner and be referred to tissue viability for a static or deteriorating wound

Exclusion Criteria:

* Patients with circumferential leg ulcers

Patients with deep narrow sinus where the opening is less than 10mm

Wounds on the face where the image would include the eyes or distinguishing features

Patients unable to provide written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
comparative consistency of the image | 1 week
  comparative reliability and consistency of the image between 2d and 3d images
comparative consistency of the measurement | 1 week
  comparative reliability and consistency of the measurements between 2d and 3d images

CONTACTS AND LOCATIONS:
Overall Officials: Brenda King, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided